CLINICAL TRIAL: NCT03455868
Title: Bone Health After Bariatric Surgery in Patients With Type 2 Diabetes
Acronym: BODI
Status: Recruiting | Type: Observational
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Claudia Gagnon, Dr, CHU de Quebec-Universite Laval
Other Study IDs: MP-10-2018-2957
Record Dates: First submitted 2018-02-19; First posted 2018-03-07 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery; Bone Health; Obesity, Morbid; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2 | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (serum and plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sleeve gastrectomy diabetes: 70 Men and women with or without type 2 diabetes and obesity undergoing sleeve gastrectomy
  Interventions: Procedure: Bariatric surgery
- Control without obesity or diabetes: 30 Men and women who are overweight (without obesity) and without diabetes

INTERVENTIONS:
Procedure: Bariatric surgery — Sleeve gastrectomy
  Groups: Sleeve gastrectomy diabetes

SUMMARY:
Background: Bone fragility is a complication of type 2 diabetes. Diabetes treatments may ameliorate or deteriorate bone fragility in this population. Bariatric surgery is gaining in popularity in people with type 2 diabetes and may impact bone health. Objectives: To evaluate the impact of the most popular bariatric procedure worldwide (sleeve gastrectomy (SG)) on vBMD by QCT in patients with type 2 diabetes; Secondary aims: (1) to identify the determinants of vBMD after bariatric surgery in patients with type 2 diabetes; (2) to compare vBMD and its potential determinants after bariatric surgery with obese controls without diabetes as well as with controls without obesity and normoglycemia.

DETAILED DESCRIPTION:
This is a multicentre, prospective and observational study comprising a bariatric group with or without diabetes undergoing SG (n=70) and one control group (n=30).

Outcome measures are assessed before and at 4 months, 8 months, one year and 3 years after surgery in the bariatric groups and at a single visit for the control group.

Bariatric groups will include adult men and women with or without type 2 diabetes and obesity undergoing sleeve gastrectomy and followed at 0, 4 months, 8 months, 1 year and 3 years after surgery, and the control group will consist of 30 overweight individuals (10 men, 10 premenopausal women, 10 menopausal women) and without diabetes or prediabetes and assessed at a single visit.

ELIGIBILITY:
Inclusion Criteria:

* bariatric groups: men and women; 18 to 60 years old; with a BMI >=35 kg/m2; with type 2 diabetes: use of oral hypoglycemic agents or insulin OR 2 of the following tests confirming type 2 diabetes: HbA1c >=6.5%; fasting glucose >=7.0 mM; 2-h glucose post 75g oral glucose tolerance test (OGTT) >=11.1 mM) (guidelines.diabetes.ca);) or without diabetes: HbA1c <6.5% AND fasting glucose <7.0 mM; who are awaiting bariatric surgery. Control group: BMI 25.0 to 29.9 kg/m2 (overweight group); without diabetes or prediabetes: HbA1c <6.0% AND fasting glucose <6.1 mM (Diabetes Canada criteria), with a stable weight for the last 3 months.

Exclusion Criteria:

* bariatric groups: type 1 diabetes; disease (e.g. uncontrolled thyroid disease, malabsorptive or overt inflammatory disorder, metabolic bone disease, creatinine clearance <60 ml/min) or medication (e.g. glucocorticoids, anti-epileptic drugs, osteoporosis therapy and thiazolidinediones) affecting bone metabolism; BMI>60 kg/m2; CT scan impossible to perform (e.g. patient too large for the gantry aperture); pregnant women or women who plan to become pregnant during the study or women of childbearing age who do not agree to take an appropriate contraceptive method during the study; history of oesophageal, gastric or digestive surgery; history of bariatric surgery; cancer at risk of recurrence during the study; Prosthesis that could interfere with interpretation of imaging data; Chronic severe condition or illness precluding from participation in the project.

Control group: Same criteria plus: >5% change in weight in the last 3 months; pregnancy or lactation in the last year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This is a multicentre, prospective and observational study comprising a bariatric group with or without diabetes undergoing SG (n=70) and one control group (n=30).
  Bariatric groups will include adult men and women with or without type 2 diabetes and obesity undergoing sleeve gastrectomy and followed at 0, 4 months, 8 months, 1 year and 3 years after surgery, and the control group will consist of 30 overweight individuals (10 men, 10 premenopausal women, 10 menopausal women) and without diabetes or prediabetes and assessed at a single visit.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in volumetric bone mineral density (vBMD) at lumbar spine, hip, tibia and radius | before, 1 year after and 3 years after bariatric surgery
  assessed by quantitative computed tomography (QCT)
Change in areal bone mineral density at lumbar spine, hip and radius | before, 1 year after and 3 years after bariatric surgery
  assessed by dual-energy X-ray absorptiometry (DXA)

SECONDARY OUTCOMES:
Change in N-terminal propeptide of type 1 procollagen (P1NP) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  serum bone formation marker
Change in osteocalcin (total, gamma-carboxylated and and under-carboxylated) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  serum bone formation marker
Change in bone alkaline phosphatase | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  serum bone formation marker
Change in C-telopeptide | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  serum bone resorption marker
Change in fasting glucose | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  diabetes control
Change in HbA1c | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  diabetes control
Change in fasting insulin | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in serum 25-hydroxyvitamin D | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in parathormone (PTH) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in estradiol and estrone | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in insulin like growth factor (IGF)-1 | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in sclerostin | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in adiponectin | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in leptin | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in peptide YY (PYY) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in ghrelin | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in oxidative stress markers | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in serum advanced glycation end products (AGEs) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in Free fatty acids (FFA) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  hormones involved in bone metabolism
Change in fat and lean mass | before, 1 year after and 3 years after bariatric surgery
  body composition assessed by bioimpedance and by DXA
Change in visceral and subcutaneous adipose tissue | before, 1 year after and 3 years after bariatric surgery
  body composition assessed by computed tomography (CT)
Change in muscle mass and fat content at mid-femur | before, 1 year after and 3 years after bariatric surgery
  assessed by computed tomography (CT)
Change in upper extremity muscle strength | before, 1 year after and 3 years after bariatric surgery
  assessed by hand grip strength
Change in lower extremity muscle strength | before, 1 year after and 3 years after bariatric surgery
  assessed by knee extensor strength
Change in muscle function | before, 1 year after and 3 years after bariatric surgery
  assessed by timed up and go test
Change in physical capacity | before, 1 year after and 3 years after bariatric surgery
  assessed by 6-minute walk test
Change in balance | before and 1 year after bariatric surgery
  assessed by Fullerton Advanced Balance (FAB) Scale
Change in sociodemographic factors | before, 1 year after and 3 years after bariatric surgery
  questionnaire
Change in nutrition | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  3 web-based 24-h recalls
Change in self-reported physical activity level | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  by questionnaire
Change in measured physical activity level | before, 1 year after and 3 years after bariatric surgery
  by accelerometer
Change in gut microbiota | before, 1 year after and 3 years after bariatric surgery
  stool sample
Change in cutaneous Advanced glycation end products (AGEs) | before, 4 months after, 8 months after, 1 year after and 3 years after bariatric surgery
  skin autofluorescence

OTHER OUTCOMES:
Bone microarchitecture and metabolism | during surgery
  by iliac crest bone biopsy after tetracycline labelling using standard histomorphometry
Prevalence and incidence of vertebral fractures (by a CT scout of T4-L5) | before, 1 year after and 3 years after bariatric surgery
  Using the algorithm-based qualitative method (ABQ) and the Genant method
Prevalence and incidence of falls | before, 1 year after and 3 years after bariatric surgery
  by questionnaire
Prevalence and incidence of non-vertebral fractures | before, 1 year after and 3 years after bariatric surgery
  by questionnaire (self-reported)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, Dr, Principal Investigator — CHU de Québec - Université Laval
Locations (3):
- Canada (3):
  - The Research Institute of the McGill University Health Centre, Montreal, Quebec
  - Centre de recherche du CHU de Québec - Université Laval, Québec, Quebec
  - Centre de recherche de l'IUCPQ, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No